CLINICAL TRIAL: NCT02239276
Title: Expanded Access Use of Stiripentol in Participants With Dravet Syndrome or Epileptic Encephalopathies Associated With Sodium Channel Mutations
Brief Title: Expanded Access Use of Stiripentol in Dravet Syndrome or Sodium Channel Mutation Epileptic Encephalopathies
Status: No longer available | Type: Expanded Access
Sponsor: Cook Children's Health Care System (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-047
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Dravet Syndrome; Epileptic Encephalopathies Associated With SCN1A Mutations
Keywords: Stiripentol; Dravet syndrome; Epilepsy; Epileptic Encephalopathies
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy | interventions — stiripentol

INTERVENTIONS:
Drug: Stiripentol — The initial dose of Stiripentol will be determined by the prescribing neurologist and titrated up to an initial goal dose of 50 mg/kg/day divided into 2 to 3 doses per day. Further dose increases by 10-20 mg/kg/day increments up to a max of 100 mg/kg/day or 4000 mg total daily dose may be necessary for improved seizure control.
  Other Names: Diacomit

SUMMARY:
This is an expanded access use of Stiripentol in Dravet Syndrome or epileptic encephalopathies associated with sodium channel mutations who have failed other drugs in an effort to give them the best chance at seizure control and quality of life. As a treatment protocol and not a research study, children will only be monitored on a clinical basis for seizure improvement and side effects predominantly by parent and caregiver report.

DETAILED DESCRIPTION:
The initial dose of Stiripentol will be determined by the prescribing neurologist and titrated up to an initial goal dose of 50 mg/kg/day divided into 2 to 3 doses per day. Further dose increases by 10-20 mg/kg/day increments up to a max of 100 mg/kg/day or 4000 mg total daily dose may be necessary for improved seizure control.

Stiripentol is available as gelatin capsules and powder sachets (250 mg, 500 mg). The same granule formulation (i.e. active, PVP and portion of sodium starch glycolate) used for the capsule is used in the final powder blend with a few additional excipients. Depending upon patient weight, the 250 mg or 500 mg formulation will be utilized for each participant.

Caretakers will be queried about common adverse effects including drowsiness, tremor, ataxis, nausea, anorexia, weight loss, and emesis. Intolerable adverse effects will prompt dose reduction or withholding medication.

Monitoring of these and other potential AEs will occur during study visits and participant-initiated telephone calls throughout the study. Safety events and tolerability will be recorded as adverse events (AE) or serious adverse events (SAE).

Physical examination, weight, vital signs, and laboratory tests (cbc, complete metabolic panel, and AED levels) will be conducted at baseline and at least every 6 months and as clinically warranted.

ELIGIBILITY:
Inclusion Criteria:

* 6 months and older
* Diagnosis of Dravet Syndrome or epileptic encephalopathies associated with SCN1A mutations defined as:

  * A documented gene mutation reported to result in Dravet syndrome phenotype; OR
  * Clinical confirmation of Dravet syndrome by two pediatric neurologists; OR
  * Clinical confirmation of other epileptic encephalopathies associated with sodium channel mutations
* Failure of at least 2 therapeutic anticonvulsants (excluding Na Channel blockers) indicative of intractable seizures

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Past history of psychoses in the form of episodes of delirium
* Impaired hepatic and/or renal function, defined as creatinine >2 and/or transaminase >4xULN

Ages: 6 Months to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Scott Perry, MD, Principal Investigator — Cook Children's Health Care System
Locations (1):
- Cook Children's Medical Center, Fort Worth, Texas, United States

REFERENCES:
- See also: Cook Children's Health Care System website — http://www.cookchildrens.org/Pages/Default.aspx